CLINICAL TRIAL: NCT00593554
Title: A Phase II Trial of Haplotype Mismatched Hematopoietic Stem Cell Transplantation Using Highly Purified CD34 Cells in Patients With Hematological Malignancies
Brief Title: Phase 2 Haplotype Mismatched HSCT in Patients With Hematological Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Sherif S. Farag (Other)
Responsible Party: Sponsor-Investigator, Sherif S. Farag, Lawrence H. Einhorn Professor of Oncology, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0704-19 IUCRO-0184
Record Dates: First submitted 2008-01-04; First posted 2008-01-15 (Estimated); Results first posted 2018-04-10 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-03

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Myelodysplasia; Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Whole-Body Irradiation; Thiotepa; fludarabine; thymoglobulin; Antilymphocyte Serum; Fibroblast Growth Factor 7

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 (Active Comparator): Total body Irradiation; Thiotepa; Fludarabine; Rabbit ATG;
  Interventions: Radiation: Total Body Irradiation; Drug: Thiotepa; Drug: Fludarabine; Biological: Rabbit ATG
- 2 (Experimental): Palifermin; Total Body Irradiation; Thiotepa; Fludarabine; Rabbit ATG
  Interventions: Radiation: Total Body Irradiation; Drug: Thiotepa; Drug: Fludarabine; Biological: Rabbit ATG; Drug: Palifermin

INTERVENTIONS:
Radiation: Total Body Irradiation — 8 Gy on Day -9
Drug: Thiotepa — 5 mg/kg/d on Day -8 to -7
Drug: Fludarabine — 40 mg/m2/d on Day -6 to -3
Biological: Rabbit ATG — 2.5 mg/kg/d on Day -5 to -2
  Other Names: Antithymocyte globulin; Thymoglobulin
Drug: Palifermin — 60 ug/kg (actual body weight) on Day -9 to -7 and Day 0 to +2
  Other Names: Recombinant human keratinocyte growth factor; Kepivance
  Arms: 2

SUMMARY:
The purpose of this study is to determine if haplotype-mismatched HSCT is associated with an improvement in treatment-related mortality (TRM) rate at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically documented AML, ALL, MDS, CML, Acute myeloid leukemia (AML) with one or more of the following criteria

  * CR 1 with poor risk features
  * CR 2, or higher order CR
* Acute lymphoblastic leukemia (ALL) with one of the following criteria

  * CR 1 with poor risk features
  * CR 2, or higher order CR
* Myelodysplasia, RAEB I
* Donor has been identified
* Age ≤ 65 years.
* Performance Status 0-1.

Exclusion Criteria:

* Patients relapsing <6 months after autologous SCT are not eligible.
* Patients with active infections requiring oral or intravenous antibiotics are not eligible for enrollment until resolution of infection.
* Non-pregnant and non-nursing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-08-07 (Actual); Primary Completion 2016-08-27 (Actual); Study Completion 2017-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Farag, MD/PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Cancer Center, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This protocol had 9 enrolled patients, but one patient never received a transplant nor was randomized. There had been no efficacy or safety data entered for this patient, and they are excluded from the results.
Groups:
- Treatment Without Paliferim: Total body Irradiation; Thiotepa; Fludarabine; Rabbit ATG;
  Total Body Irradiation: 8 Gy on Day -9
  Thiotepa: 5 mg/kg/d on Day -8 to -7
  Fludarabine: 40 mg/m2/d on Day -6 to -3
  Rabbit ATG: 2.5 mg/kg/d on Day -5 to -2
- Treatment With Palifermin: Palifermin; Total Body Irradiation; Thiotepa; Fludarabine; Rabbit ATG
  Total Body Irradiation: 8 Gy on Day -9
  Thiotepa: 5 mg/kg/d on Day -8 to -7
  Fludarabine: 40 mg/m2/d on Day -6 to -3
  Rabbit ATG: 2.5 mg/kg/d on Day -5 to -2
  Palifermin: 60 ug/kg (actual body weight) on Day -9 to -7 and Day 0 to +2
Period: Overall Study
Arm/Group | Treatment Without Paliferim | Treatment With Palifermin
Started | 3 | 5
Completed | 0 | 0
Not Completed | 3 | 5
Not completed — Death | 1 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Disease Progression | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Without Paliferim | Treatment With Palifermin | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (13.73) | 45.9 (12.21) | 44.6 (11.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Treatment-related Mortality (TRM) Rate at 6 Months After Transplantation
Description: To determine if haplotype-mismatched HSCT is associated with a ≤40% treatment-related mortality (TRM) rate at 6 months after transplantation; a TRM ≥60% being considered unacceptable. The percent of patients with the exact 95% confidence interval who had treatment-related mortality within 6 months of their transplant is presented.
Time Frame: thru 6 months after transplant
Population: Patients who received a transplant
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment Without Paliferim | Treatment With Palifermin
Number analyzed (Participants) | 3 | 5
percentage of patients | 33 [0 to 91] | 0 [0 to 0]

2. Secondary Outcome: Regimen-related Toxicity
Description: The number of unique patients who had adverse events that were possibly/probably/definitely related to treatment/regimen.
Time Frame: Up to 1 year
Population: Patients who received a transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Without Paliferim | Treatment With Palifermin
Number analyzed (Participants) | 3 | 5
Participants | 0 | 0

3. Secondary Outcome: Time to Neutrophil Engraftment
Description: Time to neutrophil engraftment will be analyzed by the Kaplan-Meier method. The time to engraftment of neutrophil is defined as the time from transplant until absolute neutrophil count (ANC) > 500 uL for 3 consecutive days. The median and 95% confidence intervals will be provided.
Time Frame: Transplant (Day 0) up to 1 year
Population: Patients who received a transplant
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment Without Paliferim | Treatment With Palifermin
Number analyzed (Participants) | 3 | 5
days | 15 [11 to 23] | 14 [7 to 28]

4. Secondary Outcome: Time to Platelet Engraftment
Description: Time to platelet engraftment will be analyzed by the Kaplan-Meier method. The time to engraftment of platelets is defined as the time from day 0 to the first of seven consecutive days after transplantation during which the platelet count is at least 20 x109/l without transfusion support. Only patients who achieved engraftment of platelets will be included in the analysis. The median and 95% confidence intervals will be provided.
Time Frame: Transplant (Day 0) up to 1 year
Population: Patients who received a transplant and who achieved platelet recovery/engraftment of platelets
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment Without Paliferim | Treatment With Palifermin
Number analyzed (Participants) | 3 | 5
days | 22.5 [17 to 28] | 20 [14 to 73]

5. Secondary Outcome: Acute Graft vs. Host Disease (GvHD)
Description: Number of unique patients who had acute Graft vs. Host Disease (GvHD) diagnosed while on the study.
Time Frame: Up to 1 year
Population: Patients who received a transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Without Paliferim | Treatment With Palifermin
Number analyzed (Participants) | 3 | 5
Participants | 0 | 0

6. Secondary Outcome: Chronic Graft vs. Host Disease (GvHD)
Description: Number of unique patients who had chronic Graft vs. Host Disease (GvHD) diagnosed while on the study.
Time Frame: Up to 1 year
Population: Patients who received a transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Without Paliferim | Treatment With Palifermin
Number analyzed (Participants) | 3 | 5
Participants | 0 | 0

7. Secondary Outcome: Frequency of Infection
Description: Number of unique patients with bacterial and/or viral infections reported.
Time Frame: Day 0 through 1 year post transplantation
Population: Patients who received a transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Without Paliferim | Treatment With Palifermin
Number analyzed (Participants) | 3 | 5
Participants | 2 | 5

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Treatment Without Paliferim | Treatment With Palifermin
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/5
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Without Paliferim (N=3) | Treatment With Palifermin (N=5)
PAIN - OTHER (General disorders) | 0 | 1
INFECTION - OTHER (Infections and infestations) | 0 | 1
INFECTION WITH UNKNOWN ANC - LUNG (PNEUMONIA) (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Without Paliferim (N=3) | Treatment With Palifermin (N=5)
BLOOD/BONE MARROW - OTHER (Blood and lymphatic system disorders) | 1 | 0
COAGULATION - OTHER (Blood and lymphatic system disorders) | 1 | 0
FEBRILE NEUTROPENIA (FEVER OF UNKNOWN ORIGIN WITHOUT CLINICALLY OR MICROBIOLOGICALLY DOCUMENTED INFE (Blood and lymphatic system disorders) | 1 | 4
LYMPHATICS - OTHER (Blood and lymphatic system disorders) | 1 | 0
THROMBOTIC MICROANGIOPATHY (E.G., THROMBOTIC THROMBOCYTOPENIC PURPURA [TTP] OR HEMOLYTIC UREMIC SYND (Blood and lymphatic system disorders) | 0 | 1
CARDIAC GENERAL - OTHER (Cardiac disorders) | 0 | 1
LEFT VENTRICULAR DIASTOLIC DYSFUNCTION (Cardiac disorders) | 0 | 1
PERICARDIAL EFFUSION (NON-MALIGNANT) (Cardiac disorders) | 1 | 1
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA - ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA - SINUS TACHYCARDIA (Cardiac disorders) | 3 | 4
VENTRICULAR ARRHYTHMIA - VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 1
OCULAR/VISUAL - OTHER (Eye disorders) | 1 | 0
VISION-BLURRED VISION (Eye disorders) | 1 | 1
ASCITES (NON-MALIGNANT) (Gastrointestinal disorders) | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 2
DIARRHEA (Gastrointestinal disorders) | 3 | 5
DISTENSION/BLOATING, ABDOMINAL (Gastrointestinal disorders) | 1 | 0
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 2 | 0
ILEUS, GI (FUNCTIONAL OBSTRUCTION OF BOWEL, I.E., NEUROCONSTIPATION) (Gastrointestinal disorders) | 0 | 2
MUCOSITIS/STOMATITIS (CLINICAL EXAM) - ORAL CAVITY (Gastrointestinal disorders) | 1 | 2
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) - LARGE BOWEL (Gastrointestinal disorders) | 0 | 1
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) - ORAL CAVITY (Gastrointestinal disorders) | 2 | 2
NAUSEA (Gastrointestinal disorders) | 3 | 5
PAIN - ABDOMEN NOS (Gastrointestinal disorders) | 2 | 3
PAIN - ORAL CAVITY (Gastrointestinal disorders) | 0 | 1
PAIN - RECTUM (Gastrointestinal disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 3 | 5
CONSTITUTIONAL SYMPTOMS - OTHER (General disorders) | 0 | 1
EDEMA: LIMB (General disorders) | 3 | 5
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 3 | 5
PAIN - OTHER (General disorders) | 1 | 2
PAIN - PAIN NOS (General disorders) | 0 | 1
RIGORS/CHILLS (General disorders) | 0 | 2
BILIRUBIN (HYPERBILIRUBINEMIA) (Hepatobiliary disorders) | 3 | 4
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 1
HEPATOBILIARY/PANCREAS - OTHER (Hepatobiliary disorders) | 1 | 0
COLITIS, INFECTIOUS (E.G., CLOSTRIDIUM DIFFICILE) (Infections and infestations) | 1 | 2
INFECTION - OTHER (Infections and infestations) | 3 | 3
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - BLADDER (URINARY) (Infections and infestations) | 0 | 1
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - BLOOD (Infections and infestations) | 0 | 1
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - ORAL CAVITY-GUMS (GINGIVITIS) (Infections and infestations) | 0 | 1
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - SINUS (Infections and infestations) | 0 | 1
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - UPPER AIRWAY NOS (Infections and infestations) | 0 | 1
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - VAGINA (Infections and infestations) | 0 | 1
INFECTION WITH UNKNOWN ANC - BLADDER (URINARY) (Infections and infestations) | 0 | 3
INFECTION WITH UNKNOWN ANC - BLOOD (Infections and infestations) | 1 | 3
INFECTION WITH UNKNOWN ANC - CATHETER-RELATED (Infections and infestations) | 0 | 1
INFECTION WITH UNKNOWN ANC - COLON (Infections and infestations) | 0 | 1
INFECTION WITH UNKNOWN ANC - LIP/PERIORAL (Infections and infestations) | 0 | 1
INFECTION WITH UNKNOWN ANC - LUNG (PNEUMONIA) (Infections and infestations) | 0 | 1
INFECTION WITH UNKNOWN ANC - ORAL CAVITY-GUMS (GINGIVITIS) (Infections and infestations) | 0 | 1
INFECTION WITH UNKNOWN ANC - SINUS (Infections and infestations) | 0 | 2
INFECTION WITH UNKNOWN ANC - UPPER AIRWAY NOS (Infections and infestations) | 0 | 3
RASH: DERMATITIS ASSOCIATED WITH RADIATION - RADIATION (Injury, poisoning and procedural complications) | 0 | 1
ALKALINE PHOSPHATASE (Investigations) | 3 | 4
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Investigations) | 3 | 5
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 3 | 4
CREATININE (Investigations) | 2 | 4
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 4
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) - EXTREMITY-LOWER (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN - BACK (Musculoskeletal and connective tissue disorders) | 2 | 2
PAIN - BONE (Musculoskeletal and connective tissue disorders) | 0 | 1
PAIN - EXTREMITY-LIMB (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN - JOINT (Musculoskeletal and connective tissue disorders) | 0 | 1
PAIN - MUSCLE (Musculoskeletal and connective tissue disorders) | 0 | 2
DIZZINESS (Nervous system disorders) | 1 | 1
ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
EXTRAPYRAMIDAL/INVOLUNTARY MOVEMENT/RESTLESSNESS (Nervous system disorders) | 1 | 0
MEMORY IMPAIRMENT (Nervous system disorders) | 0 | 1
NEUROPATHY: SENSORY (Nervous system disorders) | 1 | 3
PAIN - HEAD/HEADACHE (Nervous system disorders) | 2 | 1
CONFUSION (Psychiatric disorders) | 0 | 1
INSOMNIA (Psychiatric disorders) | 0 | 1
MENTAL STATUS (Psychiatric disorders) | 0 | 2
MOOD ALTERATION - DEPRESSION (Psychiatric disorders) | 0 | 1
HEMORRHAGE, GU - BLADDER (Renal and urinary disorders) | 0 | 1
HEMORRHAGE, GU - URINARY NOS (Renal and urinary disorders) | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 1 | 0
RENAL/GENITOURINARY - OTHER (Renal and urinary disorders) | 1 | 2
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 | 1
HEMORRHAGE, GU - VAGINA (Reproductive system and breast disorders) | 0 | 1
IRREGULAR MENSES (CHANGE FROM BASELINE) (Reproductive system and breast disorders) | 0 | 1
PAIN - PERINEUM (Reproductive system and breast disorders) | 0 | 1
ADULT RESPIRATORY DISTRESS SYNDROME (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ALLERGIC RHINITIS (INCLUDING SNEEZING, NASAL STUFFINESS, POSTNASAL DRIP) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 3
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 3 | 4
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY - NOSE (Respiratory, thoracic and mediastinal disorders) | 1 | 1
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY - RESPIRATORY TRACT NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2 | 3
MUCOSITIS/STOMATITIS (CLINICAL EXAM) - PHARYNX (Respiratory, thoracic and mediastinal disorders) | 0 | 1
NASAL CAVITY/PARANASAL SINUS REACTIONS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PAIN - THROAT/PHARYNX/LARYNX (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURAL EFFUSION (NON-MALIGNANT) (Respiratory, thoracic and mediastinal disorders) | 2 | 1
PULMONARY/UPPER RESPIRATORY - OTHER (Respiratory, thoracic and mediastinal disorders) | 0 | 2
DERMATOLOGY/SKIN - OTHER (Skin and subcutaneous tissue disorders) | 1 | 0
HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 | 1
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 0 | 2
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 2 | 2
HYPERTENSION (Vascular disorders) | 0 | 1
HYPOTENSION (Vascular disorders) | 1 | 1
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes